CLINICAL TRIAL: NCT05159817
Title: Monocentre, Observational Clinical Study Evaluating the Efficacy and Safety of a Novel Interposition Supraciliary Implant in Glaucoma Surgery
Brief Title: Study of an Interposition Supraciliary Implant in Patients With Open Angle Glaucoma
Acronym: SAFARI FU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ciliatech (Industry)
Responsible Party: Sponsor
Other Study IDs: SAFARI FU
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to prolong observational follow-up up to 36 months of patients already implanted with a novel interposition supraciliary implant.

DETAILED DESCRIPTION:
19 patients with primary open angle glaucoma (POAG) refractory to topical medical therapy were operated in late 2020 and a novel interposition supraciliary device implanted.

These patients reached 6 months follow-up and the original study had to be interrupted.

This observational study prolonges follow-up to 36 months

ELIGIBILITY:
Inclusion Criteria:

* All patients who were implanted in this center with the novel supraciliary interposition device under the scope of clinical trial NCT03736655

Exclusion Criteria:

* if cannot assist to all future follow-up visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were implanted in this center with the novel supraciliary interposition device under the scope of clinical trial NCT03736655
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess post-op IOP reduction | 12, 24 and 36 months
  Proportion of Eyes With Intraocular Pressure (IOP) Reduction of ≥ 20%

CONTACTS AND LOCATIONS:
Locations (1):
- Malayan Center, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No